CLINICAL TRIAL: NCT00088114
Title: A Phase I Trial of STA-4783 in Patients Receiving Paclitaxel for Treatment of Solid Tumors
Brief Title: STA-4783 and Paclitaxel for Treatment of Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4783-01
Record Dates: First submitted 2004-07-20; First posted 2004-07-21 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

INTERVENTIONS:
Drug: STA-4783/paclitaxel

SUMMARY:
The purpose of this study is to determine the safety, toxicity and maximum tolerated dose of single doses of STA-4783/paclitaxel in combination when administered intravenously to patients with refractory cancer. To determine the pharmacokinetics of STA-4783 and paclitaxel when co-administered.

To assess the anti-tumor activity of STA-4783 and paclitaxel when co-administered.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients greater than or equal to 18 years of age with histologically confirmed malignancy that is metastatic or unresectable and for which no standard therapy exists.
* Patients must not have received prior chemotherapy or radiation for greater than or equal to 4 weeks before study enrollment.
* Patients may be entered if they have received prior radiation therapy involving less than or equal to 30% of the bone marrow. Any prior radiation therapy must have been administered greater than or equal to 4 weeks before study enrollment and the patient must be recovered from the acute toxic effects of the treatment prior to study entry.
* Patients may be enrolled with a history of treated brain metastases that are clinically stable for greater than or equal to 4 weeks prior to enrollment.
* ECOG Performance Status of less than or equal to 2.
* Life expectancy of greater than 12 weeks.
* No peripheral neuropathy > grade 1 on NCI CTC version 2 scale, no history of stroke or other significant neurological limitations as determined by the investigator.
* Patients must have acceptable organ and marrow function at screening and pre-dose visits as defined below.
* Absolute neutrophil count greater than or equal to 1,500/ul
* Platelets greater than or equal to 100,000 cells/ul
* Total bilirubin must be within normal limits
* AST(SGOT) less than or equal to 2.5 times the upper limit of normal
* Serum creatinine < 1.5 mg/dl or a measured creatine clearance greater than or equal to 50 mL/min
* Electrocardiogram without evidence of clinically significant conduction abnormalities or active ischemia as determined by investigator.
* The effects of STA-4783 on the developing human fetus are unknown, however taxanes are known to be teratogenic. Therefore, women of childbearing potential (defined as women less than or equal to 50 years of age or history of amenorrhea for < 12 months prior to study entry) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Women who are pregnant or lactating.
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients with previous high dose chemotherapy with autologous stem cell rescue bone marrow transplantation.
* Use of any investigational agents within 4 weeks of study enrollment.
* History of severe allergic reactions to paclitaxel or docetaxel including severe hypersensitivity reactions defined as greater than or equal to 3 based on NCI CTC version 2.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness/social situations that would limit compliance with study requirements, as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-01; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Beth Israel-Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts